CLINICAL TRIAL: NCT02370134
Title: Development of Parkinson's Glove for Detection and Suppression of Hand Tremor at Rest Among the Tremor-predominant Parkinson's Disease Patients With Medically Intractable Tremor
Brief Title: Development of Parkinson's Glove for Detection and Suppression of Hand Tremor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Roongroj Bhidayasiri, Comprehensive Movement Disorders Center, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 005/58
Record Dates: First submitted 2015-01-15; First posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parkinson's glove (Experimental): Parkinson's glove 14 days use with 4 times follow-up
  Interventions: Device: Parkinson's glove
- sham glove (Placebo Comparator): sham glove (with light and sound)14 days use with 4 times follow-up
  Interventions: Device: sham glove

INTERVENTIONS:
Device: Parkinson's glove — Parkinson's glove had module for detection tremor by gyroscope/acceleroscope and suppression rest hand tremor with electrical muscle stimulation
  Arms: Parkinson's glove
Device: sham glove
  Arms: sham glove

SUMMARY:
This study is aimed to study the feasibility and safety of parkinson's glove that combined 2 module of tremor detection and tremor suppression with electrical muscle stimulation for using as device for rest tremor suppression in parkinson's disease patients

DETAILED DESCRIPTION:
Study Population

1. Target: Thai Parkinson's disease (PD) patients with predominant rest tremor : 50 patients
2. Population sample: Patients who are getting their treatment at the Chulalongkorn Comprehensive Movement Disorder Clinic at King Chulalongkorn Memorial Hospital.

Study methods as follows:

* All PD subjects will be provided the information on this research study and informed consent will be sought for every subjects.
* All PD subjects will be interviewed by a movememt disorders specialist or a trained interviewer for their demographic and clinical data.
* All PD patients will be examined for the severity of Parkinson's disease by a movement disorders specialist according the Unified Parkinson's disease Rating Scale (UPDRS), Hoehn and Yahr score, and tremor rating scale during the 'on period' in order to determine the additional effect of parkinson's glove and sham glove for suppression of tremor
* All PD patients will be randomly allocated into 2 groups (25 Parkinson's glove and 25 sham glove) with block randomization method.
* All patients will get Parkinson's glove for home-based usage for 14 days, the appointment for follow -up will be done for 4 times, with once daily phone call from investigators in order to check for improvement symptoms and all adverse events such as pain will be recorded and determined it severity by the visual analog scale.

Data collection

* Demographic and clinical data: age, gender, clinical diagnosis, tremor rating scale, pain score by visual analog scale , Parkinson's disease's severity score for each subject according to establishing standard rating scale.
* Tremor parameters form Parkinson's glove will be collected in SD card as 5 parameters: Peak magnitude, RMS, Angle, Frequency, Q. Number of stimulation times will be recorded.

Data analysis The statistical analysis in this study is based from SPSS program version 17. Categorical data will be analyzed for frequency and percentage. Continuous data will be analyzed by mean and standard deviation (SD). Non-parametric study would be preferred if the small sample size or in case of distribution of data do not present as normal distribution (determined by Kolmogorov-Smirnov test). The repeated ANOVA will be used for determined the efficacy of parkinson's glove in the difference times in follow up periods.

ELIGIBILITY:
Inclusion Criteria:

* • Adults ≥ 18 years old.

  * Patients with Parkinson's disease diagnosed according to the UKPDSBB criteria with predominantly feature of rest tremor that intractable to medically treatment.
  * Informed consent

Exclusion Criteria:

* Patients with a history of cardiac arrhythmia, renal failure, hepatic failure, and pregnancy as well as those who had history of seizure or had the risk for tended to become seizure such as those who had focal brain lesions, encephalitis, and stroke patients.

  * Patients with a history of hand surgery and implanted screws or wires in hand area that supposed to place a surface EMG or EMS, as well as those patients who were implanted for electrical devices such as cardiac pacemaker, pulse generator of deep brain stimulation,and intrathecal baclofen pump.
  * Patients who cannot avoid the medication that may potentiate or attenuate tremor such as antihistamines, benzodiazepine, illicit drugs, and thyroid hormone supplement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who demonstrate the tremor suppression after use parkinson's glove | up to 1 month follow up period
  To determine the tremor suppression after use the parkinson's glove by the tremor rating scale

SECONDARY OUTCOMES:
Number of Participants who report pain or any adverse events from parkinson's glove | 14 days periods of using parkinson's glove and in subsequent 1 month follow up period
  To determine the safety of parkinson's glove
Determine the severity of pain related with parkinson's glove | 14 days periods of using parkinson's glove
  To determine the severity of pain by visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Roongroj Bhidayasiri, MD, FRCP, Study Director — Chulalongkorn University
Locations (1):
- Chulalongkorn University Hospital, Pathumwan, Bangkok, Thailand